CLINICAL TRIAL: NCT05050760
Title: An Exploratory Study of the Efficacy and Safety of DCF Regimen Combined With Camrelizumab in the Treatment of Locally Advanced Esophageal Squamous Cell Carcinoma(ESCC)
Brief Title: DCF Combined With Camrelizumab in the Treatment of Esophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: KY20212101-C-1
Record Dates: First submitted 2021-08-04; First posted 2021-09-21 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-08

CONDITIONS: ESCC
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Intervention Model Description: Patients fulfilling Eligibility Criteria will be included in our study.After three cycles of resectable esophageal cancer treated with DCF combined with camrelizumab neoadjuvant therapy, the researchers determined whether the patient should undergo surgical treatment according to clinical diagnosis and patient willingness.If the patient underwent surgery, surgery was performed 6-8 weeks after discontinuation;If the patient did not receive surgical treatment, the patient was continued to receive 3 cycles of adjuvant therapy with camrelizumab combined with DCF regimen
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The experimental group (Experimental): Drug：DCF+Camrelizumab Camrelizumab:200mg/time,IV,Q3W
  Interventions: Drug: Camrelizumab; Drug: DCF

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab 200mg IV D1，Q3W,and preoperative therapy with three cycles.
Drug: DCF — DCF:Oxaliplatin (85mg/ m^2, IV D1,Q3W.Docetaxel: 60 mg/m^2 intravenous infusion for 60 minutes, D1,Q3W.Tegafur:BSA<1.25^2,40 mg/time,1.25^2<BSA<1.5^2,50 mg/time,BID ,after breakfast and dinner, continuous administration for 14 days, rest for 7 days, as a treatment cycle;Repeat every 3 weeks

SUMMARY:
To evaluate the safety and feasibility of DCF combined with camrelizumab in the treatment of locally advanced ESCC

DETAILED DESCRIPTION:
Primary outcome:

To evaluate the safety and feasibility of DCF combined with camrelizumab in the treatment of locally advanced ESCC

Secondary outcome:

pathologic complete response (pCR)、Major Pathologic Response（MPR）、R0 resection rate、Objective response rate（ORR）、Disease free survival（DFS）、Relief rate and safety of dysphagia

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old patients with esophageal cancer, male and female.
2. A patient with esophageal squamous cell carcinoma diagnosed by pathology.
3. Initial treatment, no previous surgery.
4. Subjects were patients with resectable locally advanced ESCC(AJCC V8 TNM classification),tumor node metastasis classification(TNM)
5. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group(ECOG) Performance Scale.
6. Expected survival ≥ 3 months.
7. All patients should have measurable or evaluable target lesions.
8. Able to eat more than a liquid diet; No preesophageal perforation signs; There was no distant metastasis and the operation was tolerated.
9. Demonstrate adequate organ function.
10. Male subjects whose partners are women of childbearing age should be surgically sterilized or agree to use an effective method of contraception during the study period and for 3 months after the last study administration.
11. The subjects voluntarily joined the study and signed the informed consent, with good compliance and follow-up.

Exclusion Criteria:

1. Patients who did not meet the inclusion criteria for pathological type and primary site.
2. Known to be allergic to macromolecular protein preparations, or components of carilizumab, or to loplatin, docetaxa, sergiol, contrast agents and their preparations.
3. Risk of esophageal perforation or presence of esophageal ulcers.
4. There is evidence of distant organ metastasis.
5. Surgical treatment (except biopsy), radiotherapy, chemotherapy, and molecular targeted therapy have been performed.
6. had other malignant tumors ever.
7. History of severe lung or heart disease.
8. Active infection or fever of unknown cause > 38.5℃ in the 2 weeks prior to randomization (fever due to tumor can be included in the study as determined by the investigator).
9. Significant active infection is known, or the investigator determines the presence of significant blood, renal, metabolic, gastrointestinal, or endocrine dysfunction.
10. Have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
11. Subjects requiring systematic treatment with corticosteroids (>10mg/ day of prednisone efficacy dose) or other immunosuppressive agents within 14 days prior to the first study drug. In the absence of active autoimmune disease, inhaled or topical steroid use and adrenal corticosteroid replacement at a dose >10mg/ day of prednisone efficacy dose were permitted.
12. Participants had active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), and hepatitis C (HCV antibody positive and HCV-RNA higher than the lower limit of the assay).
13. Those who had received live vaccine within 3 months prior to treatment.
14. In the midst of acute or chronic tuberculosis infection.
15. Patients were enrolled in clinical trials of other antitumor drugs within 4 weeks.
16. IV fluids cannot be administered.
17. She has a history of gastrointestinal ulcer, gastrointestinal bleeding and perforation.
18. Have a history of gastrointestinal ulcer, gastrointestinal bleeding and perforation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Feasibility（Incidence of Treatment-Emergent Adverse Events） | 12months
  All participants with treatment-related adverse events as assessed by National Cancer Institute Common Terminology Criteria for Adverse Event,Version 5.0(CTC AE5.0).

SECONDARY OUTCOMES:
Pathologic Complete Response (PCR) | 1 month after resection
  PCR is defined as pT0N0M0
Major pathologic response (MPR) | 1 month after resection
  MPR is defined as viable tumor comprised ≤ 10% of resected tumor specimens.
Disease Free Survival (DFS) | 3 and 5 years
  Percentage of Participants With DFS, as Assessed by RECIST 1.1. DFS is defined as the time from randomization to the first documented disease progression of local recurrence or distant metastasis or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Yang, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China